CLINICAL TRIAL: NCT04775966
Title: CPAP Observance During the COVID-19 (SARS-CoV-2) Pandemic
Acronym: COVADENE
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0067
Record Dates: First submitted 2021-02-26; First posted 2021-03-01 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Sleep Apnea Syndromes
Keywords: Sleep Apnea; Positive Airway Pressure; telemedicine; COVID 19
MeSH Terms: conditions — Sleep Apnea Syndromes; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study population: Patients meeting eligibility criteria (see appropriate section).

SUMMARY:
The hypothesis of this work is that the COVID 19 pandemic and the associated lockdowns are likely to modify the adherence to positive airway pressure (PAP) treatments among patients with sleep apnea. Identifying these patients and identifying adherence "trajectories" over time would help mobilize human and telemedicine resources on the patients most in need.

DETAILED DESCRIPTION:
The primary objective of this study is to compare PAP adherence during lockdowns in 2020 with the corresponding weeks during 2019.

ELIGIBILITY:
Inclusion Criteria:

* patient treated/monitored by the Adene group
* treated for sleep apnea syndrome (i.e., an initial apnoea hypopnea index (iAHI) ≥ 30/h or iAHI ≥ 15/h (and more than 10/h respiratory-effort-related arousal or cardio-metabolic/respiratory comorbidities) associated with symptoms from among sleepiness, tiredness, snoring, headaches, hypertension, reduced vigilance, libido disorders, nocturia, choking or suffocation during sleep, daytime tiredness)
* Positive airway pressure (PAP)-treated for at least 4 months before January 1, 2019
* continuous PAP during 2019
* continuous PAP during 2020
* acceptance of PAP telemonitoring with consent given for data collection and data anonymization

Exclusion Criteria:

* less than 360 daily PAP tele-monitored data per year for 2019
* less than 360 daily PAP tele-monitored data per year for 2020

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the Adene group database treated with positive airway pressure (PAP) for sleep apnea in 2019 and 2020.
Sampling Method: Probability Sample
Enrollment: 8477 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Change in positive airway pressure(PAP)-adherence during the first lockdown versus corresponding 2019 weeks (h/days) | 2020 versus 2019

SECONDARY OUTCOMES:
Change in positive airway pressure(PAP)-adherence during the second lockdown versus corresponding 2019 weeks (h/days) | 2020 versus 2019
Change in PAP-adherence 2020 versus 2019 (h/days/weeks) | 2020 versus 2019
Change in the percentage of adherent patients (adherence > 4h/day/week) during the first lockdown versus corresponding 2019 weeks (h/days) | 2020 versus 2019
Change in the percentage of adherent patients (adherence > 4h/day/week) during the second lockdown versus corresponding 2019 weeks (h/days) | 2020 versus 2019
Change in patient adherence 2020 versus 2019 (%). | 2020 versus 2019

CONTACTS AND LOCATIONS:
Overall Officials: Dany Jaffuel, MD,PhD, Study Director — Montpellier University Hospitals
Locations (1):
- Adene Group, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bertelli F, Suehs CM, Mallet JP, Court-Fortune I, Gagnadoux F, Borel JC, Gaubert O, Molinari N, Bourdin A, Jaffuel D. Did COVID-19 impact Positive Airway Pressure adherence in 2020? A cross-sectional study of 8477 patients with sleep apnea. Respir Res. 2022 Mar 4;23(1):46. doi: 10.1186/s12931-022-01969-z. PMID 35246109